CLINICAL TRIAL: NCT06661278
Title: Evaluation of Free-living Physical Activity and the Assessment Tools Used to Support Pharmacological Therapy Titration and Exercise Prescription in Children and Adolescents Diagnosed With Inherited Arrhythmias
Brief Title: Evaluation of Exercise Testing and Physical Activity in Children and Adolescents Living With Inherited Arrhythmias
Acronym: ACTIVELY
Status: Recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Renwick Catherine, Consultant Nurse / HEE/NIHR Doctoral Clinical and Practitioner Academic Fellow, Royal Brompton & Harefield NHS Foundation Trust
Other Study IDs: 341211
Record Dates: First submitted 2024-08-29; First posted 2024-10-28 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Long QT Syndrome; Catecholaminergic Polymorphic Ventricular Tachycardia Type 1; Catecholaminergic Polymorphic Ventricular Tachycardia Type 2
Keywords: Children; Adolescents; Exercise; Physical activity; Exercise tolerance testing
MeSH Terms: conditions — Long QT Syndrome; Polymorphic Catecholaminergic Ventricular Tachycardia; Motor Activity | interventions — Exercise Test; Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected: Children diagnosed with Long QT Syndrome and Catecholaminergic Polymorphic Ventricular Tachycardia
  Interventions: Diagnostic Test: Exercise tolerance test; Other: Physical activity & heart rate monitoring
- Unaffected: Healthy children (siblings of affected or those undergoing screening)
  Interventions: Diagnostic Test: Exercise tolerance test; Other: Physical activity & heart rate monitoring

INTERVENTIONS:
Diagnostic Test: Exercise tolerance test — Clinical routine exercise tolerance test using an exercise treadmill, according to the arrhythmia protocol (15 minute protocol utilising increasing speed and incline with a 6 minute recovery)
Other: Physical activity & heart rate monitoring — Physical activity monitoring over two weeks using Actiheart and Pro-Diary monitors to record heart rate, heart rhythm, activities engaged in and estimated intensity of activities.

SUMMARY:
The goal of this observational study is to evaluate exercise testing and daily physical activity in children and adolescents who are diagnosed with an inherited arrhythmia.

The main question it aims to answer is: Does maximum heart rate during controlled exercise tolerance testing accurately reflect maximum heart rate and peak exercise levels during free living daily physical activity in children and adolescents diagnosed with an inherited arrhythmia?

Participants will:

* Complete routine exercise tolerance testing
* Record daily physical activity and exercise over two weeks, while wearing an activity and heart rate monitor and digit diary.
* Complete a physical activity questionnaire at the end of two weeks.

DETAILED DESCRIPTION:
Exercise tolerance testing (ETT) using an exercise treadmill is a tool used to assess children's physical response to stress, which is thought to accurately reflect normal physiology during normal daily activities and can be used to:

* Evaluate heart rhythm and symptoms occurring during exercise.
* Evaluate children with a family history of sudden death and inherited heart conditions.
* Assess the response of medications prescribed to control heart rhythm.

The maximum heart rate achieved during ETT is used to estimate the effect of daily medications and to guide exercise prescription.

Originally designed to assess adult heart disease patients, ETTs were not intended for use in children. To accommodate the needs of children, shorter ETT protocols have been developed which increase the speed and/or incline of the treadmill quickly.

Despite this, many children rarely complete the full ETT protocol as they grow tired or develop other symptoms, which leads to them stopping exercise early, resulting in variable lengths of testing.

Children naturally increase exercise effort during day-to-day free-living physical activity (PA). Free-living PA is therefore thought to show a more accurate representation of the maximum heart rate (HR) children can achieve. Presently there is no strong evidence base to determine what children with an Inherited Arrhythmia (IA) (a genetically inherited heart condition which causes abnormalities in the heart rhythm) are doing in terms of daily free-living PA and exercise. The current recommendations used to prescribe exercise for this patient group are based on expert opinion and are not child specific. The study I propose supports the development of a greater evidence base to guide future exercise prescription and better tailored medications.

The study aims to:

* To compare the maximum HR achieved during controlled ETT with the maximum HR achieved during daily free-living PA and exercise, to see if these are different.
* To assess three different exercise testing protocols for children, and identify if one is better than the others at estimating maximum heart rate compared with free-living PA.
* To investigate the actual versus reported PA children engage in using a questionnaire and digital PA diary.

To achieve these aims, the study will recruit children (aged 6-16 years) diagnosed with an IA and who are able to run on an exercise treadmill, plus a healthy control group (unaffected siblings, or children undergoing screening).

A clinical ETT will be performed as part of routine care. Each participant will be given a wearable PA monitoring device to monitor free-living PA over two-weeks. The device will record parameters such as electrocardiogram, HR, and step count. PA will also be recorded digitally to capture type and length of activity they engage in, and estimated intensity.

At the end of the two-weeks, participants will complete a questionnaire about their PA which will be compared with the data obtained during the monitoring period. Parents will be invited to support younger children with questionnaire and digital recording completion.

A study lay advisory group will be established including children and their parents affected by an IA. They will advise on study design and development of all patient-facing information throughout the study.

The results of the study will be discussed with lay advisory groups who will advise on the best ways to share results with the wider public but will include publication in high quality Open Access journals and dissemination at relevant national and international conferences. Invitations will also be provided to the voluntary support groups involved in the early planning phases to publish the results on their websites

ELIGIBILITY:
Inclusion Criteria:

Affected cohort

* Male and female children
* Aged 6-16 years
* Diagnosed with long QT syndrome or catecholaminergic polymorphic ventricular tachycardia
* Treated with beta-blocker and/or sodium channel blockade
* Able to complete a treadmill ETT

Healthy cohort

* Male and female children
* Aged 6-16 years
* Siblings of affected children (gene negative)
* Undergoing IAS screening
* Able to complete a treadmill ETT

Exclusion Criteria:

* Children aged less than 6 years
* Adults, 17 years of age and above
* Unable to run on an exercise treadmill due to physical limitations.
* Individuals unable to speak or understand English, due to no translation service available.
* Pregnancy

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Affected cohort: 60 children aged 6-16 years, diagnosed with inherited arrhythmias (IAS)
  Unaffected cohort: 50 healthy children aged 6-16 years (siblings of affected children and those undergoing screening for inherited arrhythmias)
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of maximum heart rate during clinical exercise tolerance test and daily physical activity | Baseline assessment (week one of study assessments)
  Assess the correlation between maximum heart rate (HRmax) obtained during controlled exercise tolerance test (ETT) and wearable heart rate devices during daily free-living (FL) physical activity (PA) and exercise.
Physical activity questionnaire | End of two-week physical activity monitoring (week two of study assessments)
  Investigate actual versus reported PA children engage in using a questionnaire to record accuracy of child/parent recall of the type and intensity of PA.

SECONDARY OUTCOMES:
Heart rate assessment during exercise tolerance testing | Baseline assessment (week one of study assessment)
  Assess differences in HRmax relative to age of children completing three ETT protocols i. Bruce/modified Bruce with accelerated sprint - Evelina London Children's Hospital (ELCH) ii. Arrhythmia high intensity (HIT) - Royal Brompton Hospital (RBH) iii. Arrhythmia - Great Ormond Street Hospital (GOSH)
Comparison of exercise tolerance testing protocols | Immediately after the intervention
  To compare protocols between the centres to determine if one protocol correlates more closely with HRmax (protocol completion or no further rise in HR despite increasing workload) achieved during FL PA.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Renwick, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - Royal Brompton Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No
To be completed

REFERENCES:
- [Background] Chockalingam P, Wilde AA. Inherited arrhythmia syndromes leading to sudden cardiac death in the young: a global update and an Indian perspective. Indian Heart J. 2014 Jan-Feb;66 Suppl 1(Suppl 1):S49-57. doi: 10.1016/j.ihj.2013.11.008. Epub 2013 Dec 17. PMID 24568830
- [Background] Zarain-Herzberg A, Estrada-Aviles R, Fragoso-Medina J. Regulation of sarco(endo)plasmic reticulum Ca2+-ATPase and calsequestrin gene expression in the heart. Can J Physiol Pharmacol. 2012 Aug;90(8):1017-28. doi: 10.1139/y2012-057. Epub 2012 Jul 11. PMID 22784385
- [Background] Gibbons RJ, Balady GJ, Beasley JW, Bricker JT, Duvernoy WF, Froelicher VF, Mark DB, Marwick TH, McCallister BD, Thompson PD, Winters WL Jr, Yanowitz FG, Ritchie JL, Cheitlin MD, Eagle KA, Gardner TJ, Garson A Jr, Lewis RP, O'Rourke RA, Ryan TJ. ACC/AHA guidelines for exercise testing: executive summary. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on Exercise Testing). Circulation. 1997 Jul 1;96(1):345-54. doi: 10.1161/01.cir.96.1.345. No abstract available. PMID 9236456
- [Background] Mellor GJ, Behr ER. Cardiac channelopathies: diagnosis and contemporary management. Heart. 2021 Jun 11;107(13):1092-1099. doi: 10.1136/heartjnl-2019-316026. No abstract available. PMID 33589428
- [Background] Cheung CC, Laksman ZW, Mellor G, Sanatani S, Krahn AD. Exercise and Inherited Arrhythmias. Can J Cardiol. 2016 Apr;32(4):452-8. doi: 10.1016/j.cjca.2016.01.007. Epub 2016 Jan 14. PMID 26927864
- [Background] Bruce RA, Blackmon JR, Jones JW, Strait G. Exercising testing in adult normal subjects and cardiac patients. 1963. Ann Noninvasive Electrocardiol. 2004 Jul;9(3):291-303. doi: 10.1111/j.1542-474X.2004.93003.x. No abstract available. PMID 15245347
- [Background] Sagray E, Allison TG, Wackel PL. Is a high-intensity exercise test better than a graded exercise test in eliciting exercise-related arrhythmias? HeartRhythm Case Rep. 2021 May 15;7(8):549-552. doi: 10.1016/j.hrcr.2021.05.001. eCollection 2021 Aug. No abstract available. PMID 34434706
- [Background] Duff DK, De Souza AM, Human DG, Potts JE, Harris KC. A novel treadmill protocol for exercise testing in children: the British Columbia Children's Hospital protocol. BMJ Open Sport Exerc Med. 2017 Apr 22;3(1):e000197. doi: 10.1136/bmjsem-2016-000197. eCollection 2017. PMID 28761700
- [Background] van der Cammen-van Zijp MH, Ijsselstijn H, Takken T, Willemsen SP, Tibboel D, Stam HJ, van den Berg-Emons RJ. Exercise testing of pre-school children using the Bruce treadmill protocol: new reference values. Eur J Appl Physiol. 2010 Jan;108(2):393-9. doi: 10.1007/s00421-009-1236-x. Epub 2009 Oct 11. PMID 19821120
- [Background] CAVAGNA GA, SAIBENE FP, MARGARIA R. MECHANICAL WORK IN RUNNING. J Appl Physiol. 1964 Mar;19:249-56. doi: 10.1152/jappl.1964.19.2.249. No abstract available. PMID 14155290
- [Background] Schepens B, Willems PA, Cavagna GA. The mechanics of running in children. J Physiol. 1998 Jun 15;509 ( Pt 3)(Pt 3):927-40. doi: 10.1111/j.1469-7793.1998.927bm.x. PMID 9596810
- [Background] Van Hooren B, Fuller JT, Buckley JD, Miller JR, Sewell K, Rao G, Barton C, Bishop C, Willy RW. Is Motorized Treadmill Running Biomechanically Comparable to Overground Running? A Systematic Review and Meta-Analysis of Cross-Over Studies. Sports Med. 2020 Apr;50(4):785-813. doi: 10.1007/s40279-019-01237-z. PMID 31802395
- [Background] Schoffl I, Ehrlich B, Stanger S, Rottermann K, Dittrich S, Schoffl V. Exercise Field Testing in Children: A New Approach for Age-Appropriate Evaluation of Cardiopulmonary Function. Pediatr Cardiol. 2020 Aug;41(6):1099-1106. doi: 10.1007/s00246-020-02359-2. Epub 2020 May 9. PMID 32388667
- [Background] Pelliccia A, Sharma S, Gati S, Back M, Borjesson M, Caselli S, Collet JP, Corrado D, Drezner JA, Halle M, Hansen D, Heidbuchel H, Myers J, Niebauer J, Papadakis M, Piepoli MF, Prescott E, Roos-Hesselink JW, Graham Stuart A, Taylor RS, Thompson PD, Tiberi M, Vanhees L, Wilhelm M; ESC Scientific Document Group. 2020 ESC Guidelines on sports cardiology and exercise in patients with cardiovascular disease. Eur Heart J. 2021 Jan 1;42(1):17-96. doi: 10.1093/eurheartj/ehaa605. No abstract available. PMID 32860412
- [Background] Priori SG, Blomstrom-Lundqvist C. 2015 European Society of Cardiology Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death summarized by co-chairs. Eur Heart J. 2015 Nov 1;36(41):2757-9. doi: 10.1093/eurheartj/ehv445. PMID 26745817
- [Background] Maron BJ, Chaitman BR, Ackerman MJ, Bayes de Luna A, Corrado D, Crosson JE, Deal BJ, Driscoll DJ, Estes NA 3rd, Araujo CG, Liang DH, Mitten MJ, Myerburg RJ, Pelliccia A, Thompson PD, Towbin JA, Van Camp SP; Working Groups of the American Heart Association Committee on Exercise, Cardiac Rehabilitation, and Prevention; Councils on Clinical Cardiology and Cardiovascular Disease in the Young. Recommendations for physical activity and recreational sports participation for young patients with genetic cardiovascular diseases. Circulation. 2004 Jun 8;109(22):2807-16. doi: 10.1161/01.CIR.0000128363.85581.E1. PMID 15184297
- [Background] Chaput JP, Willumsen J, Bull F, Chou R, Ekelund U, Firth J, Jago R, Ortega FB, Katzmarzyk PT. 2020 WHO guidelines on physical activity and sedentary behaviour for children and adolescents aged 5-17 years: summary of the evidence. Int J Behav Nutr Phys Act. 2020 Nov 26;17(1):141. doi: 10.1186/s12966-020-01037-z. PMID 33239009
- [Background] Moss AJ, Zareba W, Hall WJ, Schwartz PJ, Crampton RS, Benhorin J, Vincent GM, Locati EH, Priori SG, Napolitano C, Medina A, Zhang L, Robinson JL, Timothy K, Towbin JA, Andrews ML. Effectiveness and limitations of beta-blocker therapy in congenital long-QT syndrome. Circulation. 2000 Feb 15;101(6):616-23. doi: 10.1161/01.cir.101.6.616. PMID 10673253
- [Background] Ussher MH, Owen CG, Cook DG, Whincup PH. The relationship between physical activity, sedentary behaviour and psychological wellbeing among adolescents. Soc Psychiatry Psychiatr Epidemiol. 2007 Oct;42(10):851-6. doi: 10.1007/s00127-007-0232-x. Epub 2007 Jul 17. PMID 17639309

DOCUMENTS (1):
  • Informed Consent Form (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT06661278/ICF_000.pdf